CLINICAL TRIAL: NCT04843202
Title: Determining Guideline Adherence During the Premedication Visit
Brief Title: Clinical Guidelines in Premedication Visit
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: HIM Health Information Management GmbH (Unknown)
Responsible Party: Principal Investigator, Simone Kagerbauer, Specialist in anesthesiology, Technical University of Munich
Other Study IDs: 450/20 S-EB
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Non-cardiac Surgery; Adults
Keywords: premedication; guidelines; software

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to determine the frequency with which individual guideline recommendations on preoperative evaluation of patients scheduled for non-cardiac surgery are implemented as well as identifying the guidelines that are most frequently violated.

DETAILED DESCRIPTION:
This study is a monocentric retrospective analysis. Data are extracted from the electronic premedication protocol (premedication patient data management system, PDMS). A total of 2000 adult patients are randomly selected who were seen in the premedication outpatient clinic of Klinikum rechts der Isar between June 2018 and June 2020. The information from the premedication questionnaire will be transferred to a new premedication module. The new premedication software then outputs the appropriate guideline recommendations that would have been applicable in the particular case. Using a logic stored in this system, the current guideline recommendations of the European Society of Anaesthesiology (ESA) (De Hert, Staender et al. 2018) and the recommendations of the German Society for Anesthesiology and Intensive Care Medicine (DGAI) (Geldner 2017) that apply to the respective case are pointed out on the basis of the patient data entered, for example the recommendation to discontinue or change medication or the order of additional examinations such as pulmonary function testing or echocardiography.

By comparison with the old premedication sheet, it is determined which guideline recommendations were followed and which were not. The respective guideline recommendations and their compliance or non-compliance are transferred to a table for further evaluation. A random sample of 2000 patients will be studied.

Guideline adherence to each recommendation is determined, as well as the possible organizational reasons for not following them.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen in the outpatient clinic between June 2018 and June 2020

Exclusion Criteria:

* age<18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Random sample of all patients >18 years of age seen in the premedication outpatient clinic from June 2018 to June 2020. This restriction is made because the guidelines used in this study apply only to adult patients.
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Guideline adherence | June 2018-June2020
  Determine the frequency with which individual guideline recommendations on preoperative evaluation are implemented.

CONTACTS AND LOCATIONS:
Locations (1):
- Technical University of Munich, Munich, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available on request

REFERENCES:
- [Background] De Hert S, Staender S, Fritsch G, Hinkelbein J, Afshari A, Bettelli G, Bock M, Chew MS, Coburn M, De Robertis E, Drinhaus H, Feldheiser A, Geldner G, Lahner D, Macas A, Neuhaus C, Rauch S, Santos-Ampuero MA, Solca M, Tanha N, Traskaite V, Wagner G, Wappler F. Pre-operative evaluation of adults undergoing elective noncardiac surgery: Updated guideline from the European Society of Anaesthesiology. Eur J Anaesthesiol. 2018 Jun;35(6):407-465. doi: 10.1097/EJA.0000000000000817. PMID 29708905
- [Derived] Kagerbauer SM, Wissler J, Blobner M, Biegert F, Andonov DI, Schneider G, Podtschaske AH, Ulm B, Jungwirth B. Anaesthesiologists' guideline adherence in pre-operative evaluation: a retrospective observational study. Perioper Med (Lond). 2024 Jun 28;13(1):64. doi: 10.1186/s13741-024-00424-5. PMID 38943163